CLINICAL TRIAL: NCT02971917
Title: A Clinical Study of TRUVIEW ART(Advanced Reconstruction Tech)to Improve Image Quality on Chest Radiograph
Brief Title: A Clinical Study of TRUVIEW ART™(Advanced Reconstruction Tech)to Improve Image Quality on Chest Radiograph
Acronym: ART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin Mo Goo, Professor, Department of Radiology, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUHTruviewART-001
Record Dates: First submitted 2016-11-15; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Thoracic Diseases
Keywords: Chest radiography; Image improvements; Image Reconstruction; Preprocessing; MTF
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clinical study of TRUVIEW ART (Experimental): Chest x-ray image acquisition Creation of TRUVIEW ART applied image Comparison of TRUVIEW ART image with original image
  Interventions: Radiation: Chest x-ray image acquisition; Radiation: Creation of TRUVIEW ART applied image; Radiation: Comparison of TRUVIEW ART image with original image

INTERVENTIONS:
Radiation: Chest x-ray image acquisition — Obtain a digital X-ray chest image of the patient
Radiation: Creation of TRUVIEW ART applied image — Application of TRUVIEW ART to the original chest x-ray image to create a new set of TRUVIEW ART applied image.
  Outcome: 2 versions of chest image
  1. Original Chest X-ray (w/o TRUVIEW ART)
  2. TRUVIEW ART applied image
Radiation: Comparison of TRUVIEW ART image with original image — Comparison of 2 versions of chest image side by side Performance evaluation may consist of detailed categories such as expression of chest structure, visibility level of pulmonary vascular system, etc. For all categories visibility and preference will be scored and each category will be analyzed to point out any statistical difference

SUMMARY:
To validate the following theory: "With TRUVIEW ART™ applied a detector's quantitative performance index, MTF(Modulation Transfer Function), is increased 20% or more". This is to examine the effect of the increased MTF index, whether it influences or not the interpreter's preference

DETAILED DESCRIPTION:
Background of Study :

DRTECH Corp. has developed and applied for patenting the unique technology of TRUVIEW ART™. TRUVIEW ART™ is advanced image reconstruction technology that restores image quality from the side effects of scattering signals in indirect type scintillator detectors. It is an advanced image pre-processing technology that constructs signal scattering models (PSF) of indirect type detector scintillators. Image sharpness (MTF) is improved by predicting scattering models and eliminating the scattering signal.

Purpose of Research and Assumption :

Indirect conversion type detectors using scintillators are universal in today's diagnostic imaging area. However, they have a disadvantage of signal scattering compared with direct conversion type detectors. TRUVIEW ART™(Advanced Reconstruction Technology) can restore images from the scattering problems. The purpose of this study is to verify how well it improves the usefulness in clinical diagnostic imaging. Evaluation will measure the improvements in MTF, which is the quantitative performance index of a detector.

ELIGIBILITY:
Inclusion Criteria:

* Adults of age 20 or higher
* Person who is able to fully understand the clinical research procedures
* Signed up agreement form
* Patient who visits for Chest computed tomography (CT)

Exclusion Criteria:

* Subject is pregnant or suspicious of being pregnant
* Not able or willing to provide Informed Consent, or consent is withdrawn
* Not able to collect all required case information

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Qualitative research using Wilcoxon's signed rank test to compare images produced by test equipment before and after applying TRUVIEW ART (Advanced Reconstruction Tech) | Report composed based on analysis of clinical images accumulated over 6 months
  - Preference score : Eleven anatomic regions(unobscured lung, hilum, minor fissure, retrocardiac lung, lung projected below the diaphragm (subdiaphragmatic lung), azygoesophageal recess, heart border, rib, proximal airway, thoracic spine, and overall appearance) are evaluated. Each pair of images is ranked on a scale from one to five

CONTACTS AND LOCATIONS:
Overall Officials: Jin Mo Goo, M.D., Principal Investigator — Department of Radiology, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes